CLINICAL TRIAL: NCT03150472
Title: Safety and Efficacy Evaluation of the Ivory Dentin Graft Device
Acronym: IvoryGraft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivory Graft Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QF-04-09-01P
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Deficiency of Alveolar Ridge (Disorder); Alveolar Bone Grafting; Mandibular Prosthesis User
Keywords: Dental Instruments; Dental Technology

STUDY DESIGN:
Intervention Model Description: The Ivory Dentin Graft study is a prospective, randomized, semi double blinded with blinded assessments study comparing patients grafted with Ivory Dentin Graft (study arm) and patients grafted with OsteoBiol Gen Os (control arm) for alveolar ridge preservation following tooth extraction.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the graft performing sub-investigator and the study coordinator will be un-blinded to the patient allocation. All efforts and measures would be taken by the study team to keep the patient and blinded assessors blinded of allocation (allocation of each extracted site) - semi double blinded study.
  Shipment tubes for biopsy (primary endpoint) are labelled with the appropriate blinded coded specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivory Dentin Graft (Ivory Graft Ltd.) (Experimental): Ivory Dentin Graft is a bone graft material for the repair or augmentation of bone defects in dental procedures. It consists of sterile 300 - 1200 μm porous particles or granules of hydroxyapatite which retain the natural form of the source porcine dentin and also the natural protein matrix which consists largely of porcine collagen.
  This type of Graft Matrix will be administered as the intervention.
  Interventions: Device: Graft Matrix
- OsteoBiol Gen-Os ® (Tecnoss) (Active Comparator): A natural replicate of autologous bone, Gen-Os® conserves the same intimate structures (matrix and porous form) and presents a highly osteoconductive properties.
  It is biocompatible and bioavailable, as recognized by tests made according to the ISO 10993 method conducted at Eurofins Biolab.
  This type of Graft Matrix will be administered as the intervention.
  Interventions: Device: Graft Matrix

INTERVENTIONS:
Device: Graft Matrix — Both Graft matrix products are supplied sterile, for single use only and packed in vials or a syringe-like applicator. All products consist of the same bone graft particles with the only variants being due to different amounts per package or different containers.

SUMMARY:
Ivory Dentin Graft is at least as good as the competitor treatment group (OsteoBiol Gen Os) for alveolar ridge preservation following tooth extraction.

The non-inferiority endpoints will be achieved if the competitor treatment group will not be statistically better than the Ivory Graft treatment.

DETAILED DESCRIPTION:
Device Description - Investigational Medicinal Product Ivory Dentin Graft is a bone graft material for the repair or augmentation of bone defects in dental procedures. It consists of sterile 300 - 900 μm porous particles of hydroxyapatite which retain the natural form of the source porcine dentin.

Ivory Dentin Graft is intended to be used as a bone graft material for the repair or augmentation of bone defects in dental procedures.

OsteoBiol Gen Os. - Comparator control device A natural replicate of autologous bone, Gen-Os® conserves the same intimate structures (matrix and porous form) and presents a highly osteoconductive properties. Gen-Os® is gradually resorbable and provides support in bone neoformation helping to preserve the original graft shape and volume.

Study Design: The Ivory Dentin Graft study is a prospective, randomized, semi double blinded with blinded assessments study comparing patients grafted with Ivory Dentin Graft (Investigational group) and patients grafted with OsteoBiol Gen Os (comparator group) for alveolar ridge preservation following tooth extraction.

Study Population and Justification: A total of 44 adult patients in 2 study groups scheduled to undergo at least one dental implant placement of mandibular premolar or molar are planned to be enrolled. The patients will be randomized into two treatment groups: One group is to be grafted with Ivory Dentin Graft while the second group will be grafted with OsteoBiol Gen Os, randomization ratio of 1:1 between the experimental and control group.

Sample size Justification and Statistical Analysis Plan: The rationale for sample size calculation is based on demonstrating non-inferiority in the study primary endpoint between the tested and the reference treatment groups.

The calculations assume a difference of up to 30% (percent as in unit of measure and not of relative difference) woven bone between the treatments, which will be considered equivalent (non-inferiority) and standard deviation of 32%.

In a sample of 15 patients per group, a difference of up to 30% in the mean woven bone between the treatment groups will be considered equivalent with 5% significance level and 80% statistical power. Assuming expected dropout rate of ~30%, 44 patients (22 per group) will be recruited in order to ensure final sample size of 30 study completers (15 per group). All tests will be two-tailed, and a p value of 5% or less will be considered statistically significant. The data will be analysed using the R version 4.0.1 (R development Core Team. Vienna, Austria).

Primary Endpoints: 95% Confidence Interval of the Differences between the treatments (Mean Ivory Graft - Mean Comparator) in woven bone ratio at 4 months after grafting will be applied. The non-inferiority endpoint will be achieved if the lower limit of the confidence interval will be higher than -30 (meaning that the comparator is less than 30 points better than Ivory Graft or not better at all).

Secondary Endpoints: Differences in categorical secondary endpoints will be tested for significance using Chi-Square test or Fisher's Exact test (as appropriate) Differences in numeric secondary endpoints will be tested for significance using the two-sample T-test or Non-parametric Wilcoxon-Mann-Whitney Rank sum test for independent samples (as is appropriate).

Exploratory Endpoints: Usability, defined as ease of procedure using 10-points satisfaction scale, will be summarized in appropriate tables by treatment.

The percent of teeth which require additional grafting at implant placement will be summarized and compared using Chi-square test or Fisher's exact test (as is appropriate).

Handling of Participant Withdrawals: Participants who leave the study prematurely will be replaced. A patient discontinuing the study before grafting of Ivory Dentin Graft (Visit 2) will be followed for safety. Each case of premature withdrawal will be properly recorded in the Screening Failure Log as deemed necessary.

Patient Screening: Prior to any study-related screening procedure, delegated study team members will approach potentially eligible adult patients who are waiting to be scheduled for tooth extraction and grafting for necessary titanium implant placement. Patients who do not meet inclusion criteria or who are for any other reason determined to be unsuitable for inclusion in the study, or who decline to participate in the study, will be considered and recorded as "screening failure" and receive standard and appropriate treatment.

Informed Consent: The informed consent document will be signed and dated for screening and enrollment and each patient consenting will be documented in the patient medical binder. The patient will be given a copy of the consent form together with the study doctor's letter at the time of enrollment. The clinician will ask the patient about his plans and his willingness to attend all scheduled follow-up visits.

Randomization will be done by Castor EDC web-software. The patients will be randomized into two treatment groups: One group is to be grafted with Ivory Dentin Graft while the second group will be grafted with OsteoBiol Gen Os, randomization ratio of 1:1 between the experimental and control group.

TRIAL PROCEDURES: After informed consent is obtained, a case record form including all aspects listed below will be recorded. Eligible patients will be enrolled into the study and be treated according to standard treatment protocols for tooth extraction, grafting, implant placement, dental biopsy and dental radiographic procedures and with the standard protocol for local anesthetic.

Visit 1: Screening and Enrolment, as part of pre-operative visit (0-90 days before grafting procedure ) The following assessments will be performed: Demographics, Medical history, Vital signs, Current medications. A CT scan will be performed in order to verify patient eligibility and graft procedure preparation Visit 2: Randomization and extraction socket graft filling by Ivory Dentin Graft or Gen Os after tooth extraction.

The designated randomization groups (Ivory Dentin Group and Gen Os) will be:

1. Recorded in the patient CRF
2. A sticker of the used study item and the used package will be achived in the patient binder- this will be used as source to verify correct allocation.

All patients will be operated by study delegated physicians using the same method.

Socket debridement and cleaning: After exposure of the defect the sounding walls should be debrided by surgical curette and all granulation tissue removed.

The extraction site will be graft filled either using Ivory Dentin Graft or OsteoBiol Gen-Os according to the respective Instructions for Use using either vial or syringe applicators with dental membrane. Only the graft performing sub-investigator and the study coordinator will be un-blinded to the patient allocation. All efforts and measures would be taken by the study team to keep the patient and blinded assessors blinded of allocation- semi double blinded study.

Periapical x-ray imaging will be performed on each enrolled patient once completing the graft filling in order to validate the bone grafting procedure.

The following assessments will be performed following the procedure:

1. Extraction socket grafting Physician usability Form
2. Study Patient Discharge form. Patients will be monitored for short-term follow-up (1 week, 1 and 4 months following their extraction socket grafting procedure) and for long-term follow-up and will be evaluated for their medical and dental conditions. Implantation of titanium implants will be conducted 4 months following the grafting procedure at grafted site of each enrolled patient.

Short-term Visit 3: Follow up 1 week following grafting procedure The patient will be asked to report any dental complication- all will be investigated by the sub-investigator using Visit 3 safety Follow Up Form. In addition, vital signs will be taken by study investigator.

Visit 4: Follow up 1 month following grafting procedure The patient will be asked to report any dental complication- all will be investigated by the sub-investigator using Visit 4 safety Follow Up Form. In addition, vital signs will be taken by study investigator.

A Computerized Tomography (CT) will be performed prior to visit 5 Visit 5: Follow up 4 months following grafting procedure and dental Implant placement (Short-term Termination visit)

Prior to the procedure, the patient will be asked to report any dental complication. The following assessments will be conducted during the visit:

1. Vital Signs
2. Implant placement Physician usability Form
3. Study Patient Discharge form.
4. Short-term termination visit The alveolar bone strength (torque measurement) will be measured by torque measurement.

Adequacy of bone graft (need for additional grafting at implant placement) will be evaluated by the study investigator based on the clinical examination, torque measurement and CT scan, and will be specified and justified in the Case Report Form.

Un-scheduled visit: The study investigator will instruct the patient to immediately contact the study team in case of: Implant failure, loose graft particles, loss of grafting material, graft site infection, insufficient healing of graft site, excessive bleeding and wound dehiscence. The patient must call the study nurse to schedule an un-scheduled visit which may only be performed by the principal Investigator.

Post-Market Clinical Follow-up: Patients will be monitored also for long-term follow-up (6 and 10 months, 2.5 and 5 years following their extraction socket grafting procedure) and will be evaluated by the study nurse for their medical and dental conditions.

Data Monitoring and Quality Control:The investigator, through an appointed Clinical Research Associate (CRA), will be responsible for implementing and maintaining quality assurance and quality control systems with written Standard Of Procedures to ensure that trials are conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirement(s), including ISO 14155.

The investigator will be responsible for ensuring direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the hospital, and inspection by Israeli regulatory authorities.

Quality control should be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly.

The study CRA will verify that (a) The rights and well-being of human patients are protected, (b) The reported trial data are accurate, complete, and verifiable from source documents and (c) The conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with the applicable regulatory requirement(s) (including ISO 14155). The full responsibilities of the trial monitor appear in full in the ICH-GCP. The monitor(s) should follow Ivory Graft (or their CRO representative) written for monitoring the specific trial. The monitor will submit a written report after each trial-site visit or trial-related communication. A report should include the date, site, name of the monitor, and name of the investigator or other individual(s) contacted. A report should include a summary of what the monitor reviewed and the monitor's statements concerning the significant findings/facts, deviations and deficiencies, conclusions, actions taken or to be taken and/or actions recommended to secure compliance.

To ensure compliance of this investigator initiated trial with current national regulations and the ICH guidelines, data generated by this study will be available for inspection upon request by representatives of the local health authorities- IRB or the national authorities - MOH, or any entity providing support for this trial. Routine monitoring or audit activities for this study will be conducted by authorized representatives. The general scope of such visits would be to inspect study data (regulatory requirements), source documentation and CRF completion in accordance with current GCP, the ICH guidelines and the respective local and national government regulations and guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient 18 up to 80 years.
2. Patient requiring at least one implant placement following mandibular pre-molar or molar tooth extraction.
3. Alveolar mandibular ridge (empty socket):

   * Height: not less than 10 mm, from the gingival margin to the mandibular nerve canal - as seen in the screening CT scan.
   * Width: not less than 5 mm, from buccal to lingual cortical plates - as seen in the screening CT scan.
4. Ability to give informed consent for the study by patient or legal guardian.
5. Willingness to undergo all follow up visits, as well as unscheduled sick visits.

   Exclusion Criteria:
6. Pregnancy (all women of child-bearing age would be questioned and told by the consenting physician regarding that criteria).
7. Known or suspected hypersensitivity to the constituents of the bone graft material (for example porcine collagen)
8. Pathologies or conditions contraindicating surgery or presenting with active acute or chronic infections excluding periapical granuloma (for example osteomyelitis, sinusitis), uncontrolled diabetes
9. Immunologic disorders or auto-immune pathologies, in particular elderly
10. Serious bone diseases of endocrine aetiology
11. Serious disturbances of bone metabolism
12. Ongoing treatment with gluco- or mineralocorticoids, or with agents affecting calcium metabolism (e.g. calcitonin, bisphosphonates)
13. Irradiation therapy, chemotherapy or immunosuppressive therapy in the last 5 years
14. Malignancies
15. Severe Parafunction (bruxism and clenching)
16. Poor oral hygiene or active periodontitis
17. Heavy tobacco smoking habit (> 10 cigarettes per day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Amount of new bone formation | 4 months after grafting
  Mean area of mineralized and non-mineralized tissue in alveolar bone core biopsies - "woven bone" (Ratio 0-100%)
Bone-Graft material integration score to host bone in the alveolar bone core | 4 months after grafting
  1 - poor: no signs of new bone-to-graft interface visible, 2 - intermediate: minimal and focal signs of new- bone-to-graft interface visible, 3 - good: abundant new bone-to-graft interface visible.

SECONDARY OUTCOMES:
Alveolar bone strength | 4 months after grafting
  torque measurement, comparison of Ivory Dentin Graft sites with the comparator, Gen Os.
Alveolar bone radiodensity (Hounsfield scale) | 4 months after bone grafting
  calculated by volumetric CT imaging
Success of dental implant placement in a rigid post bone grafting site | 4 months after bone grafting
  defined by immediate dental implant stability
Changes from baseline in alveolar bone height (depth reduction) | 4 months after bone grafting
  measured at mesial and distal root surface [in millimetres] on Posterior to Anterior (PA) radiographs or by computer tomography (CT).
Changes from baseline in alveolar bone width (horizontal bone gain or loss) | 4 months after bone grafting
  [in millimetres] on Posterior to Anterior (PA) radiographs or by computer tomography (CT)

OTHER OUTCOMES:
Usability study measures | at bone grafting visit and 4 months from bone grafting
  defined by the ease of the graft/implant placement procedure (scored by the physician performing the procedure using the 10-point satisfaction scale)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Lavi, PhD, Study Director — Ivory Graft Ltd.
Locations (1):
- Assaf HaRofeh Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not intended to be shared as this will be a single site study. The study will be public at ClinicalTrial.gov

REFERENCES:
- [Background] Abraham CM. A brief historical perspective on dental implants, their surface coatings and treatments. Open Dent J. 2014 May 16;8:50-5. doi: 10.2174/1874210601408010050. eCollection 2014. PMID 24894638
- [Background] Atieh MA, Alsabeeha NH, Payne AG, Duncan W, Faggion CM, Esposito M. Interventions for replacing missing teeth: alveolar ridge preservation techniques for dental implant site development. Cochrane Database Syst Rev. 2015 May 28;2015(5):CD010176. doi: 10.1002/14651858.CD010176.pub2. PMID 26020735
- [Background] Binderman I, Hallel G, Nardy C, Yaffe A, Sapoznikov L. A novel procedure to process extracted teeth for immediate grafting of autogenous dentin. J Interdiscipl Med Dent Sci, 2014; 2(6). http://dx.doi.org/10.4172/jimds.1000154
- [Background] Campbell KM, Casas MJ, Kenny DJ. Ankylosis of traumatized permanent incisors: pathogenesis and current approaches to diagnosis and management. J Can Dent Assoc. 2005 Nov;71(10):763-8. PMID 16324230
- [Background] Nguyen TT, Mui B, Mehrabzadeh M, Chea Y, Chaudhry Z, Chaudhry K, Tran SD. Regeneration of tissues of the oral complex: current clinical trends and research advances. J Can Dent Assoc. 2013;79:d1. PMID 23522126
- [Background] Patel K, Mardas N, Donos N. Radiographic and clinical outcomes of implants placed in ridge preserved sites: a 12-month post-loading follow-up. Clin Oral Implants Res. 2013 Jun;24(6):599-605. doi: 10.1111/j.1600-0501.2012.02500.x. Epub 2012 Jun 3. PMID 22672611
- [Derived] Sapoznikov L, Haim D, Zavan B, Scortecci G, Humphrey MF. A novel porcine dentin-derived bone graft material provides effective site stability for implant placement after tooth extraction: a randomized controlled clinical trial. Clin Oral Investig. 2023 Jun;27(6):2899-2911. doi: 10.1007/s00784-023-04888-5. Epub 2023 Feb 24. PMID 36826514